CLINICAL TRIAL: NCT05387382
Title: Effects of Bariatric Surgery on Different Compositions of Trunk Fat and Mechanisms
Status: Completed | Type: Observational
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: kuaiI 22091
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-05

CONDITIONS: Bariatric Surgery Candidate; Adiposity; Fat Redistribution
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Plasma for estimates of metabolism indicators
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients pending bariatric surgery: A continuous cohort of patients pending bariatric surgery

SUMMARY:
This is a prospective, single-center, observational study to explore effects of bariatric surgery on different compositions of trunk fat and mechanisms.

DETAILED DESCRIPTION:
This is a prospective, single-center, observational study to explore effects of bariatric surgery on different compositions of trunk fat and mechanisms. The primary outcome is effects of bariatric surgery on different compositions of trunk fat evaluated with MRI for patients pending bariatric surgery before and 3 months after surgery. The secondary outcome is the associations of trunk fat reduction with improvement in metabolism indicators. Before patients are enrolled in this observational study, the researchers will do a detailed screening of the subjects based on the inclusion criteria and the exclusion criteria to determine if the patients are appropriate for the study. Patients who meet the conditions of the study will be required to sign an informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* BMI of >27.5 kg/m2 with T2DM;
* BMI of >32.5 kg/m2 with or without metabolic syndrome;
* Age 18-65 years old;
* T2DM duration < 15 years.

Exclusion Criteria:

* Previous history of pancreatitis or pancreatic surgery;
* Serious T2DM complications or organic diseases;
* Alcohol addiction;
* Uncontrolled mental illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients pending bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Subcutaneous Fat Area at 3 months after bariatric surgery | Baseline and 3 months after sugery
  Change from baseline subcutaneous fat area (unite in cm3) evaluated with MRI at 3 months after bariatric surgery.
Change from Baseline Visceral Fat Area at 3 months after bariatric surgery | Baseline and 3 months after sugery
  Change from baseline visceral fat area (unite in cm3) evaluated with MRI at 3 months after bariatric surgery.
Change from Baseline Liver Fat Percentage at 3 months after bariatric surgery | Baseline and 3 months after sugery
  Change from baseline liver fat percentage (unite in %) evaluated with MRI at 3 months after bariatric surgery.
Change from Baseline Pancreatic Fat Percentage at 3 months after bariatric surgery | Baseline and 3 months after sugery
  Change from baseline pancreatic fat percentage (unite in %) evaluated with MRI at 3 months after bariatric surgery.

SECONDARY OUTCOMES:
Correlation coefficient of trunk fat change with change in metabolism indicators | Baseline and 3 months after sugery
  Correlation coefficient of trunk fat changes with changes in metabolism indicators.
  1. Trunk fat changes included changes from baseline subcutaneous fat area (unite in cm3), visceral fat area (unite in cm3), liver fat percentage (unite in %), pancreatic fat percentage (unite in %) evaluated with MRI at 3 months after bariatric surgery.
  2. Changes in metabolism indicators included changes from baseline Fasting plasma glucose (unite in mmol/L), Glycated hemoglobin (unite in %), Fasting insulin (unite in uU/mL), Fasting C-peptide (unite in ng/mL), Homeostatic Model Assessment of Insulin Resistance, Low-Density Lipoprotein Cholesterol (unite in mmol/L), High-Density Lipoprotein Cholesterol (unite in mmol/L), Cholesterol (unite in mmol/L), Triglyceride (unite in mmol/L).
  3. We used Pearson Correlation Analysis to calculate the correlation coefficient of trunk fat changes with changes in metabolism indicators.

OTHER OUTCOMES:
Age | Baseline
  Age of participants (unite in year)
Gender | Baseline
  Gender of participants
Duration of Type 2 diabetes | Baseline
  Duration of Type 2 diabetes of participants (unite in year)
Number of medicine use | Baseline and 3 months after sugery
  Number of medicine use of participants
Weight | Baseline and 3 months after sugery
  Weight of participants (unite in kg)
Body mass index | Baseline and 3 months after sugery
  Body mass index of participants (unite in kg/m2)
Waist circumference | Baseline and 3 months after sugery
  Waist circumference of participants (unite in cm)
Hip circumference | Baseline and 3 months after sugery
  Hip circumference of participants (unite in cm)
Fasting plasma glucose | Baseline and 3 months after sugery
  Fasting plasma glucose of participants (unite in mmol/L)
Glycated hemoglobin |glycosylated hemoglobin | Baseline and 3 months after sugery
  Glycated hemoglobin |glycosylated hemoglobin of participants (unite in %)
Fasting insulin | Baseline and 3 months after sugery
  Fasting insulin of participants (unite in uU/mL)
Fasting C-peptide | Baseline and 3 months after sugery
  Fasting C-peptide of participants (unite in ng/mL)
Homeostatic Model Assessment of Insulin Resistance | Baseline and 3 months after sugery
  Homeostatic Model Assessment of Insulin Resistance of participants
Low-Density Lipoprotein Cholesterol | Baseline and 3 months after sugery
  Low-Density Lipoprotein Cholesterol of participants (unite in mmol/L)
High-Density Lipoprotein Cholesterol | Baseline and 3 months after sugery
  High-Density Lipoprotein Cholesterol of participants (unite in mmol/L)
Cholesterol | Baseline and 3 months after sugery
  Cholesterol of participants (unite in mmol/L)
Triglyceride | Baseline and 3 months after sugery
  Triglyceride of participants (unite in mmol/L)
Subcutaneous Fat Area | Baseline and 3 months after sugery
  Subcutaneous Fat Area of participants evaluated with MRI (unite in cm3)
Visceral Fat Area | Baseline and 3 months after sugery
  Visceral Fat Area of participants evaluated with MRI (unite in cm3)
Liver Fat Percentage | Baseline and 3 months after sugery
  Liver Fat Percentage of participants evaluated with MRI (unite in %)
Pancreatic Fat Percentage | Baseline and 3 months after sugery
  Pancreatic Fat Percentage of participants evaluated with MRI (unite in %)

CONTACTS AND LOCATIONS:
Overall Officials: Shaihong Zhu, M.D., Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

REFERENCES:
- [Derived] Cui B, Duan J, Zhu L, Wang G, Sun X, Su Z, Liao Y, Yi B, Li P, Li W, Song Z, Li Z, Tang H, Rong P, Zhu S. Effect of laparoscopic sleeve gastrectomy on mobilization of site-specific body adipose depots: a prospective cohort study. Int J Surg. 2023 Oct 1;109(10):3013-3020. doi: 10.1097/JS9.0000000000000573. PMID 37352520